CLINICAL TRIAL: NCT00146458
Title: A Phase III Randomized Trial of FDG-PET in the Management of Advanced Cervical Cancer With Enlarged Pelvic Lymph Node on MRI Image
Brief Title: Usefulness of FDG-PET for Advanced Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTRP024; NSC 92-2314-B-182A-084
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; FDG-PET; Lymph node metastasis; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Lymphatic Metastasis

INTERVENTIONS:
Procedure: 18F-fluorodeoxyglucose positron emission tomography

SUMMARY:
The objective of this study is to determinate whether the adding of FDG-PET is helpful in the treatment of advanced cervical cancer with concurrent chemoradiation.

DETAILED DESCRIPTION:
Concurrent radiotherapy and chemotherapy is the standard treatment for locally advanced cervical cancer. The radiation field should be adjusted according to the extension of disease, especially the presence of metastatic lymph nodes. At present, CT/ MRI have been applied for the detection of enlarged lymph nodes, as the reference of radiation field. However, not infrequently, a small-sized lymph node on CT/MRI may be metastatic while an enlarged node may be resulted from reactive hyperplasia.

Unlike CT/ MRI, 18F-FDG positron emission tomography (FDG-PET) provides a novel means of imaging malignancy and could differentiate benign tumor from malignancy by functional assessment. Recent studies demonstrated higher accuracy of FDG-PET scan for the evaluation of metastasis in patients with several types of cancers when compared with CT scan or MRI. But, only a few reports concerned the usefulness of FDG-PET in cervical carcinoma.

Our hypothesis is that adding FGD-PET study to a thorough MRI can provide better staging, especially on the identification of metastatic pelvic or para-aortic lymph nodes. In addition, this whole body scan may also detect occult distant metastases that are not detectable by standard workup. Our initial result of a phase II study---"A Preliminary Report of Using FDG-PET to Detect Extra-pelvic Lesions in Cervical Cancer Patients with Enlarged Pelvic Lymph Nodes Shown on MRI/CT Images" indicated that FDG-PET helped to detect occult or small metastatic lesions, and resulted in a change of radiation treatment plan. Nevertheless, for high-risk group patients, distant metastasis still occurred in a short period after treatment. Therefore, it is also our question that whether the enhancement of detection provided by FDG-PET can be translated into improvement of final overall survival.

To answer these questions, the Gynecologic Oncology Study Group in Chang Gung Memorial Hospital has designed a phase III clinical study. Patients with enlarged pelvic lymph node detected on MRI imaging are enrolled and randomized into two groups before the initiation of concurrent chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cervical cancer clinical stage FIGO I -IVA
* Histologically proven cervical carcinoma (including histologic types of squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma, adenoid cystic carcinoma, lymphoepithelial-like carcinoma and malignant mixed mullerian tumor)
* Presence of at least one enlarged pelvic lymph node (>=1.0 cm in its maximal dimension), or group of small pelvic nodes (size <1 cm), and without suspicious para-aortic lymph node metastasis or any lesion outside the pelvis by conventional MRI or CT study
* Karnofsky performance scale >=60
* Available for concurrent chemoradiation therapy of curative intent

Exclusion Criteria:

* Cervical tumor with histologic diagnosis of verrucous carcinoma or small cell carcinoma
* Other serious illness or medical condition which would interfere with extended field irradiation or chemotherapy
* Past or current history of malignancy, except for curatively treated non-melanoma skin cancer
* Patients not suitable to receive PET study either by technical or psychological reasons
* Patients who are judged to be noncompliant to treatment or not accessible for follow up

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2002-01; Study Completion 2007-12

PRIMARY OUTCOMES:
The difference of disease-free-survival and overall-survival with/ without FDG-PET at two years after treatment

SECONDARY OUTCOMES:
The incidence of additional extra-pelvic tumor metastasis detected by FDG-PET study, and its influence on the design of appropriate radiotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Sheng Tsai, M.D., Principal Investigator — Department of Radiation Oncology, Chang Gung Memorial Hospital; Tin-Chang Chang, M.D., MPH., Study Director — Director of Division of Gynecologic Oncology, Chang Gung Memorial Hospital, Linkou Medical Center; Chyong-Huey Lai, M.D., Study Chair — Chairman of Department of Obstetrics and Gynecology, Chang Gung Memorial Hospital, Linkou Medical Center
Locations (1):
- Department of Radiation Oncology, Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Result] Tsai CS, Chang TC, Lai CH, Tsai CC, Ng KK, Hsueh S, Yen TC, Hong JH. Preliminary report of using FDG-PET to detect extrapelvic lesions in cervical cancer patients with enlarged pelvic lymph nodes on MRI/CT. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1506-12. doi: 10.1016/j.ijrobp.2003.09.013. PMID 15050330